CLINICAL TRIAL: NCT05657717
Title: Otological Safety Profile of 100% Manuka Honey Application in Tympanoplasty: A Double-blinded Randomized Controlled Trial
Brief Title: Safety Profile of Applied 100% Manuka Honey in Tympanoplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21040426
Record Dates: First submitted 2022-12-02; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Chronic Suppurative Otitis Media; Tympanic Membrane; Wound
Keywords: Chronic Suppurative Otitis Media; Manuka Honey; Tympanic Membrane; Otologic Safety
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Manukamed - 100% sterile manuka honey
  Interventions: Drug: Manukamed - Manukapli 100% sterile honey wound dressing - Premium medical grade 16+ Leptospermum Scoparium New Zealand honey
- Control (No Intervention): No intervention was given. Participants receive standard wound care of the tympanic membrane which includes 0.3% Ofloxacin otic ear drops which were used twice a day for 5 days.

INTERVENTIONS:
Drug: Manukamed - Manukapli 100% sterile honey wound dressing - Premium medical grade 16+ Leptospermum Scoparium New Zealand honey — After surgical reconstruction of the tympanic membrane by grafting, Manukamed - Manukapli 100% Sterile honey wound dressing is applied onto the gelfoam to close the area, followed by an antibiotic tampon.
  Other Names: Manukamed - Manukapli 100% sterile honey wound dressing
  Arms: Intervention

SUMMARY:
Throughout history, honey has been recognized for its healing properties. The use of honey for its medicinal properties dates back to 2200 BCE.

The purpose of this clinical trial is to learn about the otological safety of 100% Medical grade Manuka Honey given to tympanoplasty patients

The main question it aims to answer is: Can 100% Medical Grade Manuka Honey given at the time of Tympanoplasty otologically safe?

Participants in the intervention group will receive a wound dressing of 100% medical grade Manuka honey after reconstructive surgery of the tympanic membrane.

Researchers will compare the intervention group to the control group assess otological safety.

DETAILED DESCRIPTION:
The aim of the present study is to conduct a randomized clinical trial to evaluate the otological safety of 100% medical grade Manuka honey on the tympanic membrane post Tympanoplasty compared to the control group. The investigation will involve 64 participants with Chronic Suppurative Otitis Media of the mucosal type, who will be randomly put into two groups (intervention or control), where the intervention group will receive a dressing of 100% sterile Manuka honey during surgery. Results of this study will inform practitioners as to the otological safety of 100% sterile Manuka honey on the tympanic membrane.

ELIGIBILITY:
Inclusion Criteria:

* Participants of 18 - 45 years of age.
* Participants with Chronic Suppurative Otitis Media of the mucosal type.
* Provision of signed and dated informed consent form. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Participants who previously received surgical therapy for Chronic Suppurative Otitis Media or have recurrent or residual disease.
* Participants with anatomical pathology results showing and/or suspecting a tumor.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of Ototoxicity - BERA | Time Frame: 5 weeks (35 days following surgery)
  Hearing function will be evaluated by conducting a Brain Evoked Response Audiometry (BERA) exam. If the BERA results show decreased stimulus of more than 10 decibels compared to baseline, treatment is started immediately.
Evaluation of Ototoxicity - Audiometry | Time Frame: 6 weeks (42 days following surgery)
  Hearing function will be evaluated by conducting a Pure Tone Audiometry exam. Results are compared to baseline and evaluated. If there is a 20db or greater decrease in pure-tone threshold at one frequency or 10db or greater decreased at 2 adjacent frequencies, treatment is started immediately.

SECONDARY OUTCOMES:
Evaluation of Ototoxicity - Symptoms - Tinnitus | Time Frame: 6 weeks (42 days following surgery)
  Participants will be asked to complete a questionnaire regarding tinnitus. Subjective symptoms are measured using a visual analog scale ranging from 1-10, with higher scores indicating worse symptoms.
Evaluation of Ototoxicity - Symptoms - Hearing Loss | Time Frame: 6 weeks (42 days following surgery)
  Participants will be asked to complete a questionnaire regarding hearing loss. Subjective symptoms are measured using a visual analog scale ranging from 1-10, with higher scores indicating worse symptoms.
Evaluation of Ototoxicity - Symptoms - Dysequilibrium | Time Frame: 6 weeks (42 days following surgery)
  Participants will be asked to complete a questionnaire regarding dysequilibrium. Subjective symptoms are measured using a visual analog scale ranging from 1-10, with higher scores indicating worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Harim Priyono, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (1):
- Faculty of Medicine - University of Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
If requested, data records without identifying patient information can be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available not more than 6 months after study completion date

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT05657717/Prot_SAP_000.pdf